CLINICAL TRIAL: NCT07164768
Title: Cognitive Function and Mental Health in Children and Youth With Type 1 Diabetes (T1D) and Its Determinants
Brief Title: Cognitive Function and Mental Health in Children and Youth With Type 1 Diabetes (T1D)
Acronym: DMBCOG
Status: Enrolling by invitation | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, DEPUTY DIRECTOR, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: JCDC/BHR/24/034
Record Dates: First submitted 2024-12-06; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Type 1 diabetes; children; cognitive function; behavioral and emotional problems; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Aliquots of serum at -80°C for measurement of Human-BDNF.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and youth with type 1 diabetes (T1D) and their parents: The Hirabai Cowasji Jehangir Medical Research Institute (HCJMRI), Pune is a Center of Excellence in type 1 diabetes and has vast experience in studying prospective cohorts with good follow up rates. It also has a registry of more than 800 children with type 1 diabetes with systematic assessment of their glycemic control and micro and macrovascular complications due to type 1 diabetes. We would like to propose a cross sectional, observational, case control study in children with T1D and healthy controls of age 10-21 years (who give assent and parents give consent; children no neurodevelopmental disorders will be enrolled in the study) from similar socio-economic class as the children with diabetes. Approximate period of enrollment will be from July 2023 to July 2025. We expect to recruit one in two of participant with type 1 diabetes from our cohort and age gender matched healthy controls without type 1 diabetes.

SUMMARY:
The Hirabai Cowasji Jehangir Medical Research Institute (HCJMRI), Pune, a Center of Excellence in type 1 diabetes (T1D), has extensive experience in studying prospective cohorts with high follow-up rates. HCJMRI maintains a registry of over 800 children with T1D, systematically assessing their glycemic control and diabetes-related complications.

Given the high prevalence of T1D in India and the lack of studies on Indian children with T1D, the investigators aim to investigate cognitive function and mental health in children and youth with T1D compared to healthy controls, exploring key determinants of these outcomes.

The investigators propose a cross-sectional, observational, case-control study involving children and youth aged 10-21 years with T1D and age- and gender-matched healthy controls from similar socio-economic backgrounds. Participants will be enrolled between July 2023 and July 2025, with assent from children and consent from parents. Those with neurodevelopmental disorders will be excluded. The investigators plan to recruit one in two eligible participants with T1D from our existing cohort, with a total sample size of 396 participants (264 cases and 132 controls), adequately powered to detect group differences with a moderate effect size.

Data on T1D exposure will be extracted from ongoing cohort records. Outcomes assessed in both groups include:

1. Cognitive functions - assessed using age-appropriate tests.
2. Behavioral and emotional problems - evaluated in children, adolescents, and young adults.
3. Quality of life - assessed using standardized tools. Potential confounders such as age, gender, socio-economic status, parental education, occupation, participant's education, and pubertal status will be considered. Random blood samples will be collected at the time of cognitive testing to measure plasma glucose, HbA1c, and Human-BDNF levels, examining associations between glycemic control and cognitive outcomes. Additionally, annual checkup data will be used to explore the impact of T1D complications on cognitive function.

Group differences in outcomes will be analyzed using ANCOVA while controlling for covariates. Regression models will assess cognitive function as a function of T1D exposure, adjusting for mediators and modifiers.

This will be one of the first studies in India to systematically examine multiple cognitive domains in a large T1D sample across a broad age range (10-21 years). Findings will enhance understanding of T1D's impact on cognitive development in an Indian context, where undernutrition is common, and T1D prevalence is rising.

Keywords: Type 1 diabetes, children, cognitive function, behavioral and emotional problems, quality of life.

DETAILED DESCRIPTION:
Objectives of the project:

1. To assess cognitive function in children with T1D in comparison with healthy controls and its determinants (parental education and occupation, parenting style and mental health of parents)
2. To study the association of parental education and occupation, parenting style and mental health of parents with child's glycemic control in children with T1D
3. To assess the stress, anxiety and depression in children, adolescents and young adults with T1D (10-21 years) in comparison with healthy controls and its impact on their quality of life
4. Methodology:

Study Subjects:

The 'Sweetlings' programme which is a charity clinic that provides holistic care to underprivileged children and youth with Type 1 Diabetes Mellitus (T1D). Currently, the clinic supports 548 children and youth with T1DM aged 0 to 22 years in the Pune region of the Western Indian State of Maharashtra.

The investigator have 382 children between 6-18 years of age and 103 who are between 18-22 years of age. Siblings of these T1D children will be included as healthy age matched controls for participation in this study. This will ensure about the age matching and also their socioeconomic status and family environment will be similar.

Sample size estimations:

The investigator expects to recruit one in two of participant with type 1 diabetes from our cohort and age gender matched healthy controls without type 1 diabetes. Sample size estimation suggests a sample size of 396 participants (264 cases and 132 controls) would be adequately powered to detect group differences with moderate effect size.

Procedure:

Institutional ethics committee approval will be obtained for the study. Children with T1D will be approached for participation and information about the study will be provided. T1D children and their parents will be recruited after obtaining informed parental consent from children less than 12 years and parent consent and child's assent for those above 12 years of age. Informed consent will be obtained from those above 18 years of age.

Exposures:

Systematic assessments of the exposures (Type 1 diabetes, Birth weight, parental education, occupation, mental health, parenting style) will be performed in the cohort. This data of recruited subjects will be extracted from available records as well as collecting their current information using a standardized questionnaire.

Glucose values and HbA1c measured in the clinic at the time of neurocognitive testing will be taken to study the associations between the glycemic control in T1D children and their neurocognitive outcomes.

Additionally, Brain Derived Neurotrophic Factor (BDNF) which is a key molecule involved in neuroplastic changes related to learning and memory will also be measured.

Outcomes:

Cognitive function and mental health of children, adolescents and young adults with T1D Following measurements will be performed in T1D children based on their age at assessment.

1. Neurocognitive measurements: Global measures of intelligence was assessed using the Raven's progressive Matrices.
2. Mental health in children and parents: Depression, anxiety and stress related information will be collected using specific questionnaires.
3. Quality of life in children and parents using Peds QL standardised modules and questionnaires.

Cognitive function assessments (general intellectual test, IQ):

1. Raven's Colored Progressive Matrices: Raven's Progressive Matrices (often referred to simply as Raven's Matrices) or RPM is a non-verbal test typically used to measure general human intelligence and abstract reasoning and is regarded as a non-verbal estimate of fluid intelligence.
2. Speed: Finger tapping: It is the measure of motor speed. Age range: 9 years and above The finger-tapping test consists of an especially adopted electric finger-tapping instrument and monitor to read the number of taps.
3. Attention: d2: It is a refinement of the cancellation test. Age range 9-60 years.
4. Executive functioning:

   * Verbal fluency: FAS test. Age range: Children: 5 to 15 years
   * Animal names test: Age range: Children: 5 to 15 years
   * COWA test (Controlled Oral Word Association test). Adults: 15 to 65 years
   * Working memory: Digit and letter number (WISC). Age range: 6 to 16 years.
   * Processing speed: Coding and symbol search (WISC). Age range: 6 to 16 years.
   * Working memory: Digit and arithmetic (WAIS) [8] and Coding and symbol search (WAIS). Age range: 16 to 90 years
   * Working Memory Index- subtests include Digit span and arithmetic. Processing Speed Index- subtests include symbol search, coding, and cancellation.
   * Shift of set (Wisconsin card sorting test 64: Age range: 6 years 5 months to 89 years
   * Response inhibition: Stroop test. Age range: Children: 5-14 years, Adults: 15 years and above
5. Verbal learning and memory: Auditory verbal learning test (AVLT): Age range: Children: 5 to 15 years, Adults: 16 to 65 years
6. Test of comprehension: Token test: Age range: Children: 5 to 15 years, Adults: 16 to 65 years

Mental health and quality of life in children and parents:

1. CBCL (The Child Behavior Checklist): The 2001 revision of the CBCL, the CBCL/6-18 (used with children 6 to 18), is made up of eight syndrome scales:

   * anxious/depressed
   * depressed
   * somatic complaints
   * social problems
   * thought problems
   * attention problems
   * rule-breaking behaviour
   * aggressive behaviour
2. BSI (Brief Symptom Inventory): The Brief Symptom Inventory (BSI) consists of 53 items covering nine symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. The global indices measure current or past level of symptomatology, intensity of symptoms, and number of reported symptoms, respectively.
3. Quality of life:

Peds QL: The Pediatric Quality of Life Inventory (PedsQL): PedsQL Generic Core Scale will be used to measure generic health-related quality of life of the children, adolescents and young adults in this study. This scale is applicable for healthy school and community populations, as well as patient populations with acute and chronic health conditions.

Effect modifiers:

1. Parents' mental health: This will be assessed using BSI questionnaire.
2. Parenting style: The Parenting Styles and Dimensions Questionnaire (PSDQ)[19] is one measure that is widely utilized in current research to examine parenting styles.
3. Parents' quality of life: PedsQL Generic Core Scale will be used to measure generic health-related quality of life of the primary caregiver (any one parent, either mother or father).
4. Parental education and occupation: This information will be collected using standard questionnaires for general information.
5. Scholastic performance: Academic exposure can positively impact cognitive functioning. This will be assessed by taking the average marks/grades obtained by the child in previous year academic performance.

Mediators:

1. Glycemic control and complications of type 1 diabetes:

   The investigators regularly perform the annual checkups in our type 1 cohort. In that following measurements are performed to assess their glycemic control and development of micro and macrovascular complications.
2. Human BDNF (Brain Derived Neurotrophic Factor): This will be measured using standard enzymatic method using Elabscience® Human BDNF (Brain Derived Neurotrophic Factor) ELISA Kit. Association between BDNF levels and cognitive functions will be studied.
3. Growth and development: This data will be utilized from the anthropometric measurements performed at the time of their annual check-ups. Pubertal staging is performed by a pediatric endocrinologist or a medical officer. Information regarding age and date of menarche is also collected.
4. Lifestyle (nutrition and physical activity): The investigators also collect the information regarding their nutritional intake using a 24-hour dietary recall and data regarding their physical activity levels using standard questionnaire. Using this data, the investigators can study the association between lifestyle with cognitive functions

Measurement of potential confounders:

1. A semistructured proforma will be designed to collect socio-demographic information, current educational status, Parental education. Socio-economic status will be assessed using the Kuppuswamy 2023 coding and scale.
2. Family history of neurodevelopmental/neurological/mental health disorders will be obtained on a three generation genogram.
3. Pubertal status will be assessed on the Tanner's staging for Puberty by medical officer.

Future implications:

Early detection and intervention for cognitive impairment in the early stages of Type 1 Diabetes Mellitus (T1DM) can facilitate effective treatment. Cognitive impairment is closely linked to poor glycaemic control and associated metabolic disruptions in T1DM. Initiating the management of metabolic abnormalities during the initial phases of diabetes holds the potential to prevent cognitive impairment. It is essential to include cognitive impairment screening for individuals with T1DM alongside assessments for other recognised macro- and microvascular complications of diabetes.

In addition to evaluating children with T1D, conducting assessments for their parents, including an analysis of parenting styles and stress levels associated with managing their child's diabetes, allows for the strategic planning of interventions.

This holistic approach not only enhances parents' diabetes management but also contributes to improved glycaemic control in T1D children, thereby positively influencing their cognitive function.

Detecting and addressing cognitive impairment at an early stage not only aids in the effective management of diabetes in children but also plays a pivotal role in fostering improved career prospects and job opportunities for them. Additionally, this proactive approach contributes to an overall enhancement of their quality of life. The downstream effect of these positive outcomes includes a reduction in the health-related and economic burden faced by India.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and young adults with T1D and their parents (caregiver, either mother or father)

Exclusion Criteria:

* Both parents are not alive or the child is not living with the parents and living with the grandparents.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study Subjects:
  The Hirabai Cowasji Jehangir Medical Research Institute, which is a sister concern of Jehangir hospital, Pune, has been involved in health related programs since its inception in 1995. Our major areas of work include Nutritional and Growth Disorders in Children, Type 1 Diabetes, Maternal and Child Health, Osteoporosis and Bone Health, Psychological Counseling, HIV and Cancers.
  Cases: There are 738 children registered with HCJMRI for the treatment and management of type 1 diabetes. The 'Sweetlings' programme is a charity clinic that provides holistic care to underprivileged children and youth with Type 1 Diabetes Mellitus (T1D). Currently, the clinic supports 548 children and youth with T1D aged 0 to 22 years in the Pune region of the Western Indian State of Maharashtra.
  From these, we have 386 children who are between 10-21 years of age.
  Controls: Siblings of these T1D children will be included as healthy age-matched controls for participation in this study. This wil
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
To assess intelligent quotient (IQ) as a cognitive function in children and youth with type 1 diabetes | 3 years
  Age range: 4 to 90 years. Raven's Colored Progressive Matrices: Raven's Progressive Matrices (often referred to simply as Raven's Matrices) to measure general human intelligence and abstract reasoning and is regarded as a non-verbal estimate of fluid intelligence. The Raven's 2 is a nonverbal assessment of general cognitive ability, including the ability to formulate new concepts when faced with novel information, extract meaning out of confusion or ambiguity, and think clearly about complex situation and events. It comprises 60 multiple-choice questions, listed in order of increasing difficulty. This format is designed to measure the test taker's reasoning ability, the eductive ("meaning-making") component of Spearman's g (g is often referred to as general intelligence). It is a measure of verbal and nonverbal generalized cognitive ability.
To assess speed as a cognitive function in children and youth with type 1 diabetes | 3 years
  Finger-Tapping Test Age Range: 9 years and above Procedure: The test uses an adapted electric finger-tapping instrument and monitor to record the number of taps. The participant taps a mounted key as rapidly as possible using the index finger of the dominant hand, followed by the non-dominant hand. Five consecutive 10-second trials are conducted for each hand. A 30-second break is given after the third trial to minimize fatigue. A practice trial is provided before the test begins.
  Scoring: The number of taps per 10-second trial is recorded separately for each hand. The mean number of taps across five trials is calculated for each hand.
  Material: Finger-tapping instrument and stopwatch Duration: 5 minutes
To assess attention as a cognitive function in children and youth with type 1 diabetes | 3 years
  d2 Test of Attention Age Range: 9-60 years Procedure: The d2 test assesses selective attention and concentration. It can be administered individually or in groups using a single test form. The form includes sections for subject data, test scores, and a practice sample. The standardized test consists of 14 lines, each with 47 characters (total: 658 items). Participants scan each line and cross out all "d's" with two dashes. Each line is timed for 20 seconds.
  Reliability & Validity: The test demonstrates high reliability (r > 0.90) across various indices (TN, TN-E, CP) and is supported by extensive research.
  Materials: 2 pencils (without erasers) and a stopwatch for the examiner. Duration: 10 minutes
To assess phonemic fluency as an executive function in children with type 1 diabetes | 3 years
  FAS Test (Children: 5-15 years) - A phonemic fluency test measuring verbal fluency. Participants generate words beginning with F, A, and S (or Ka, Pa, Ma for non-English speakers) within one minute per letter. Proper nouns are excluded. Score: Total admissible words. Duration: ~5 minutes
To assess category fluency as an executive function in children with type 1 diabetes | 3 years
  Animal Names Test (Children: 5-15 years) - A category fluency test where participants list as many animal names as possible in one minute, excluding fish, birds, and snakes. Score: Total unique words. Duration: ~5 minutes
To assess phonemic fluency as an executive function in adolescents and youth with type 1 diabetes | 3 years
  COWA Test (Adults: 15-65 years) - A phonemic fluency test where participants generate words beginning with F, A, and S (or Ka, Pa, Ma). Proper nouns and repeated words with different suffixes are excluded. Score: Average new words over three trials. Duration: ~5 minutes
To assess category fluency as an executive function in adolescents and youth with type 1 diabetes | 3 years
  Category Fluency: Animal Names Test (Adults: 15-65 years) - Same as the children's version, assessing category fluency. Score: Total unique words. Duration: ~5 minutes
To assess working memory as an executive function in children with type 1 diabetes | 3 years
  Digit & Letter-Number (WISC) and Processing Speed: Coding & Symbol Search (WISC) Age Range: 6-16 years Developed in 2003, this scale assesses intellectual ability. The Working Memory Index (WMI) includes Digit Span, Letter-Number Sequencing, and Arithmetic (supplemental). The Processing Speed Index (PSI) includes Coding, Symbol Search, and Cancellation (supplemental).
  Digit Span: The child repeats numbers in the same or reverse order. Letter-Number Sequencing: The child recalls numbers in ascending and letters in alphabetical order.
  Symbol Search: The child scans a group to identify target symbols within a time limit.
  Duration: 10 minutes
To assess working memory as an executive function in adolescents and youth with type 1 diabetes | 3 years
  Working Memory & Processing Speed (WAIS) Age Range: 16-90 years The WMI measures working memory, attention, concentration, and reasoning, while the PSI assesses the ability to scan, sequence, and process visual information quickly. Both indices involve cognitive decision-making beyond simple reaction time.
  Duration: 20 minutes
To assess Shift of set (Wisconsin card sorting test) as an executive function in children and youth with type 1 | 3 years
  Wisconsin Card Sorting Test (WCST-64)
  Age Range: 6 years 5 months to 89 years
  The WCST-64 assesses abstract reasoning and executive functions, including cognitive flexibility, goal-directed behavior, planning, and impulse control. Unlike the full WCST, which uses 128 cards, the WCST-64 uses 64 cards. Participants match stimulus cards without explicit instructions, receiving feedback on correctness. The test generates psychometric scores on categories achieved, trials, errors, and perseverative errors.
  Materials: Four stimulus cards, 64 response cards, and a record form.
  Duration: 20-30 minutes
  The WCST has demonstrated reliability and validity across various populations, including individuals with autism, stroke survivors, pediatric groups, and psychiatric patients.
To assess Response inhibition as an executive function in children and youth with type 1 diabetes | 3 years
  Stroop Test
  Age Range: Children (5-14 years), Adults (15+ years)
  The Stroop Test measures response inhibition, assessing the ability to suppress habitual responses in favor of unusual ones. It evaluates cognitive flexibility and prefrontal function.
  Participants are shown a sheet with color names ("Blue," "Green," "Red") printed in different ink colors. They first read the words column-wise as quickly as possible while the time is recorded. Next, they name the ink color instead of reading the word, with the time again recorded.
  Score: The Stroop effect score is calculated as:
  Stroop Effect Score = Time to name colors - Time to read words Uncorrected errors are recorded separately for both phases.
  Duration: ~20 minutes
To assess Verbal Learning and Memory as cognitive function in children and youth with type 1 diabetes | 3 years
  Verbal Learning & Memory: Auditory Verbal Learning Test (AVLT)
  Age Range: Children (5-15 years), Adults (16-65 years)
  The AVLT assesses verbal learning and memory using word lists. Adapted by WHO for different cultures, it includes Lists A & B with 15 familiar words each, translated into Kannada, Tamil, Telugu, and Hindi.
  Words from List A are presented at a rate of one per second for five trials, with recall recorded after each trial. Then, List B is introduced as an interference task, followed by immediate recall of List A. After 20 minutes, delayed recall of List A is assessed without re-presentation. Finally, a recognition test is conducted by mixing List A words with new words, recording hits and errors. Words are presented in the participant's preferred language (mother tongue or English).
  Duration: 15 minutes
To assess Test of comprehension as cognitive function in children and youth with type 1 diabetes | 3 years
  Test of Comprehension: Token Test
  Age Range: Children (5-15 years), Adults (16-65 years)
  The Token Test assesses verbal comprehension using tokens that vary in color, size, and shape. Participants follow spoken instructions of increasing complexity. Squares and circles in two sizes and five colors are placed in a fixed arrangement. Instructions are given once per item, with up to two repetitions if needed.
  Scoring: One point is awarded for correct responses, with a 0.5-point deduction per repetition. A trial is failed if the participant does not follow instructions after two repetitions. The maximum score is 36.
  Duration: 20 minutes

SECONDARY OUTCOMES:
To assess mental health in children and youth with type 1 diabetes and their parents | 3 years
  CBCL (Child Behavior Checklist) Age Range: 6-18 years The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and detects behavioral and emotional problems in children. It is completed by parents, while the Teacher's Report Form (TRF) is completed by teachers, and the Youth Self-Report (YSR) by the child. The CBCL/6-18 includes eight syndrome scales: Anxious/Depressed, Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior. These form two higher-order factors: Internalizing and Externalizing. Responses cover the past six months.
  BSI (Brief Symptom Inventory) Age Range: 18 years and above The BSI has 53 items covering nine symptom dimensions, including Somatization, Obsession-Compulsion, Depression, Anxiety, and Psychoticism. It also includes three global indices measuring symptom severity, distress intensity, and total reported symptoms.
To assess Diabetes related stress and quality of life in children and youth with type 1 diabetes | 3 years
  The PedsQL Diabetes Module is a standardized tool designed to assess diabetes-related quality of life in children and adolescents with diabetes. It evaluates the impact of diabetes on various aspects of daily life, including treatment barriers, adherence, worry, and communication with healthcare providers. The module is structured for self-report by children and proxy-report by parents, covering emotional, social, and physical challenges associated with diabetes management. By identifying specific areas of distress and difficulty, the PedsQL Diabetes Module helps healthcare professionals tailor interventions to improve both medical outcomes and overall well-being in pediatric diabetes patients.
To assess parents' perception towards diabetes related stress and quality of life in their children | 3 years
  Diabetes related stress and quality of life in children and parents' perception towards quality of life in their children will be assessed using standard questionnaires developed by The PedsQL™ Diabetes Module is a specific module of the PedsQL™
To assess general quality of life in children and youth with type 1 diabetes | 3 years
  PedsQL Generic Core Scale will be used to measure generic health-related quality of life of the children, adolescnts and young adults in this study. This scale is applicable for healthy school and community populations, as well as patient populations with acute and chronic health conditions.
To assess general quality of life in parents of children and youth with type 1 diabetes | 3 years
  PedsQL Generic Core Scale[18] will be used to measure generic health-related quality of life of the primary caregiver (any one parent, either mother or father). This scale is applicable for healthy school and community populations, as well as patient populations with acute and chronic health conditions.
  4. Parental education and occupation: This information will be collected using standard questionnaires for general information.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sonali S Wagle, M.Sc, RD, PhD, Study Chair — Hirabai Cowasji Jehangir Medical Research Institute, Pune, India
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) will be shared with qualified researchers.
  The shared data will include [specify data types, e.g., demographics, clinical outcomes, etc.].
  Access will be granted to researchers with a scientifically sound proposal that has been reviewed and approved by an independent review board. Requests should be directed to [provide contact information or system, e.g., "via email to the principal investigator, Dr. Anuradha Khadilkar]. Data sharing will comply with applicable laws, regulations, and institutional policies to ensure privacy and data security.
Supporting Information: Study Protocol
Time Frame: The data will become available 6 months after publication in a scientific journal and will remain accessible for the specified period decided by the principal investigator.
Access Criteria: Access will be granted to researchers with a scientifically sound proposal that has been reviewed and approved by an independent review board. Requests should be directed to the principal investigator, Dr. Anuradha Khadilkar via email.